CLINICAL TRIAL: NCT01016652
Title: Clinical Evaluation of a Multifocal Contact Lens on Symptomatic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Collaborators: Visioncare Research Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CR-4558; VMFL-511 (Other: Visioncare Research, Ltd.)
Record Dates: First submitted 2009-11-18; First posted 2009-11-19 (Estimated); Results first posted 2014-01-23 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2017-08

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- etafilcon A multifocal / etafilcon A sphere (Other): period 1: etafilcon A multifocal worn, period 2: etafilcon A sphere worn.
  Interventions: Device: etafilcon A multifocal contact lens; Device: etafilcon A Contact Lens
- etafilcon A sphere / etafilcon A multifocal (Other): period 1: etafilcon A sphere worn, period 2: etafilcon A multifocal worn.
  Interventions: Device: etafilcon A multifocal contact lens; Device: etafilcon A Contact Lens

INTERVENTIONS:
Device: etafilcon A multifocal contact lens — low-add multifocal contact lens
Device: etafilcon A Contact Lens — standard sphere contact lens

SUMMARY:
The purpose of this study is to evaluate the effect of a multi-focal contact lens on symptomatic patients.

ELIGIBILITY:
Inclusion Criteria:

* To have signed an informed consent form (documented by the investigator in the Case Report Form [CRF]).
* Be existing daily wear spherical single-vision soft CL wearers (no extended wear in the last 3 months, but silicone hydrogels in daily wear are allowed).
* Between 35 and 47 years of age (inclusive).
* Have a CL spherical distance requirement between -1.00D and -6.00D (-6.50D refractive) in both eyes.
* Refractive astigmatism of 0.75D or less in both eyes.
* Visual symptoms associated with near vision
* Be correctable to a visual acuity of 6/9 (20/30) or better in each eye.
* Have normal eyes with no evidence of abnormality or disease. For the purpose of this study a normal eye is defined as one having:

  1. No amblyopia.
  2. No evidence of lid abnormality or infection.
  3. No conjunctival abnormality or infection.
  4. No clinically significant slit lamp findings (i.e. stromal haze, staining, scarring, Vascularization, infiltrates or abnormal opacities).
  5. No other active ocular disease.

Exclusion Criteria:

* Monovision user or multifocal CL wearer.
* Regular user of reading spectacles (i.e. daily usage).
* Requires concurrent ocular medication.
* Clinically significant (Grade 3 or 4) corneal stromal haze, corneal Vascularization, tarsal abnormalities, bulbar hyperemia, limbal hyperemia, or any other abnormality of the cornea that would contraindicate CL wear.
* Corneal staining Grade 3 in more than two regions.
* Has had any anterior ocular surgery. Has had any other ocular surgery or injury within 8 weeks immediately prior to enrollment for this study.
* Pre-existing ocular irritation that would preclude CL fitting.
* Keratoconus or other corneal irregularity.

Ages: 35 Years to 47 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2009-10-01 (Actual); Primary Completion 2009-12-01 (Actual); Study Completion 2009-12-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - North Little Rock, Arkansas
  - Blue Springs, Missouri
  - Lake Ozark, Missouri
  - Warren, Ohio
  - Kittanning, Pennsylvania
  - Warwick, Rhode Island
  - Chamberlain, South Dakota
  - Burlington, Vermont

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a four week, 49 subject, doubly-masked, daily wear, two-part crossover study. Recruited patients were emerging presbyopic (35-47 years) and soft CL wearing who were experiencing any near vision symptoms.
Pre-assignment Details: A screening questionnaire (Near Vision Questionnaire, (NVQ)) was used to recruit subjects and to provide information about the wider population.
Groups:
- Etafilcon A Multifocal/ Etafilcon A Sphere: etafilcon A multifocal/ etafilcon A sphere Arm: The first test lens for this arm, etafilcon A multifocal, was dispensed on Day 0 and to be worn a minimum of 2 hours before the assessment scheduled 12-17 days after the lens was fitted. Repeat for the second lens (sphere).
- Etafilcon A Sphere/ Etafilcon A Multifocal: etafilcon A sphere/ etafilcon A multifocal Arm: The first test lens for this arm, etafilcon A sphere, was dispensed on Day 0 and to be worn a minimum of 2 hours before the assessment scheduled 12-17 days after the lens was fitted.
  Repeat for the second lens (multifocal).
Period: Period 1
Arm/Group | Etafilcon A Multifocal/ Etafilcon A Sphere | Etafilcon A Sphere/ Etafilcon A Multifocal
Started | 25 | 24
Completed | 25 | 24
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Etafilcon A Multifocal/ Etafilcon A Sphere | Etafilcon A Sphere/ Etafilcon A Multifocal
Started | 25 (Crossover study: the completed from period 1 will crossover in period 2 to the opposite arm.) | 24 (Crossover study: the completed from period 1 will crossover in period 2 to the opposite arm.)
Completed | 25 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Etafilcon A Sphere\ Etafilcon A Multifocal: etafilcon A sphere/ etafilcon A multifocal Arm: The first test lens for this arm, etafilcon A sphere, was dispensed on Day 0 and to be worn a minimum of 2 hours before the assessment scheduled 12-17 days after the lens was fitted.
  Repeat for the second lens (multifocal).
- Total: Total of all reporting groups
Arm/Group | Etafilcon A Multifocal/ Etafilcon A Sphere | Etafilcon A Sphere\ Etafilcon A Multifocal | Total
Number analyzed (Participants) | 25 | 24 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 24 | 49
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Mean age was the same for both groups.
  years | 42.3 (3.4) | 42.3 (3.4) | 42.3 (3.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 18 | 36
  Male | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Subject Reported Overall Vision Quality Using (CLUE)TM Questionnaire
Description: The Contact Lens User Experience (CLUE) Questionnaire is a validated patient-reported outcomes questionnaire to assess patient-experience attributes of soft, disposable contact lenses in the US, ages 18-65. Scores follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response, with scores ranging from 0-120.
Time Frame: week 4
Population: Analysis was on those subjects enrolled, randomized into one of two randomized arms, and who completed the study.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Etafilcon A Multifocal: etafilcon A multifocal worn.
- Etafilcon A Sphere: etafilcon A sphere worn
Arm/Group | Etafilcon A Multifocal | Etafilcon A Sphere
Number analyzed (Participants) | 49 | 49
units on a scale | 41.0 [30.0 to 51.0] | 39.0 [28.0 to 50.0]
Statistical Analysis 1: Comparison: Etafilcon A Multifocal vs Etafilcon A Sphere; Ho: There are not significant differences between the two lenses (etafilcon A multifocal (test) vs. etafilcon A sphere (control)for Vision quality. Ha: The test lens is greater than or equal by 5 CLUE points than the control lense; Test type: Non-Inferiority or Equivalence — This is a non-inferiority analysis, with >=5 CLUE points being the non-inferiority margin; Mixed Models Analysis; Mean Difference (Final Values) = -4.14, 95% CI 2-sided [-9.86 to 1.59], Standard Error of Mean 0.12

2. Primary Outcome: Monocular Amplitude of Accommodation
Description: The amplitude of accommodation is a measure of the eyes ability to accommodate or focus on near objects. The method used was the push-up/push-down method performed monocularly. One eye was occluded and using the smallest print the subject was able to read, the reading chart was slowly moved towards the subject. The subject was asked them to indicate when the print first becomes blurred. The distance was noted and the amplitude of accommodation was calculated.
Time Frame: week 4
Population: Analysis was on those who were randomized to either treatment arm with intent to treat. One eye was chosen.
Measure: Median (Inter-Quartile Range); unit: diopters
Groups:
- Etafilcon A Multifocal: etafilcon A multifocal wearers
- Etafilcon A Sphere: etafilcon A sphere wearers
Arm/Group | Etafilcon A Multifocal | Etafilcon A Sphere
Number analyzed (Participants) | 49 | 49
diopters | 0.00 [-0.075 to 0.025] | 0.00 [-0.075 to 0.01]
Statistical Analysis 1: Comparison: Etafilcon A Multifocal vs Etafilcon A Sphere; Ho: There is not a difference between the test lens and the control lens for amplitude of accommodation. Ha: Monocular amplitude of accommodation of the test lens is significantly better than the control lens; Test type: Non-Inferiority or Equivalence — The non-inferiority margin will be exceeded if the test lens is greater than or equal to 0.25D over the control lens; Mixed Models Analysis; Mean Difference (Net) = 0.01, 95% CI 2-sided [-0.09 to 0.10], Standard Error of Mean 0.06

3. Secondary Outcome: Proportion of Subjects With Near Vision Symptoms as Assessed by the NVQ
Description: Proportion of subjects reporting frequent/constant near vision problem per the Near Vision Questionnaire (NVQ). The NVQ was used to assess subjects' near vision problems. Subjects graded each question using a 5-level Likert-type scale (5-levels: never, infrequent, sometimes, frequently, constantly).
Time Frame: week 4
Population: The NV Questionnaire was administered to those enrolled in the study and randomized to either treatment arm.
Measure: Number; unit: percentage of participants
Arm/Group | Etafilcon A Multifocal | Etafilcon A Sphere
Number analyzed (Participants) | 49 | 49
percentage of participants | 53 | 43

4. Secondary Outcome: Subject Reported Lens Comfort Using CLUE Questionnaire
Description: Subject reported lens comfort was assessed using the CLUE Questionnaire. CLUE is a validated patient-reported outcomes questionnaire to assess patient-experience attributes of soft, disposable contact lenses in the US, ages 18-65. Scores follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response. Scores range from 0 -120.
Time Frame: week 4
Population: Analysis was on those subjects enrolled and randomized to either one of the arms with intent to treat.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Etafilcon A Multifocal | Etafilcon A Sphere
Number analyzed (Participants) | 49 | 49
units on a scale | 59.0 [38.0 to 75.0] | 59.0 [50.0 to 77.0]

5. Secondary Outcome: Comfortable Wearing Time
Description: Comfortable wearing time was measured using self-reported subject awareness of irritation at a given time of day, rounded to the nearest half-hour. Could be described as aware of issue or completely comfortable.
Time Frame: week 4
Population: Analysis was on those subjects randomized to either arm with the intent to treat.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Etafilcon A Multifocal | Etafilcon A Sphere
Number analyzed (Participants) | 49 | 49
hours | 14 [11 to 15] | 14 [12 to 14.5]

6. Secondary Outcome: Proportion of Subjects Benefiting From the Binocular +/-1.00D Accommodative Flipper
Description: Utility of the use of the Binocular +/-1.00D accommodative flipper as a screening tool for those emerging presbyopia subjects
Time Frame: Baseline
Population: Analysis was on those subjects who were randomized to either treatment arm with the intent to treat.
Measure: Number; unit: percentage of participants
Arm/Group | Etafilcon A Multifocal | Etafilcon A Sphere
Number analyzed (Participants) | 49 | 49
percentage of participants | 52 | 58

ADVERSE EVENTS:
Arm/Group | Etafilcon A Multifocal | Etafilcon A Sphere
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/49
Other Adverse Events (participants affected / at risk) | 0/49 | 0/49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Written authorization by the Sponsor is required for publication.